CLINICAL TRIAL: NCT02737176
Title: Efficacy of Tobacco Cessation for Improving Oral Diseases - Multicenter Prospective Trial
Brief Title: Tobacco Cessation Intervention Study for Oral Diseases
Acronym: TISOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association for the Japanese Academy of Maxillofacial Implants (Other)
Responsible Party: Principal Investigator, Toru Nagao, PhD, DMSc, DDS, Director, Association for the Japanese Academy of Maxillofacial Implants
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssociationJAMI
Record Dates: First submitted 2016-03-31; First posted 2016-04-13 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Smoking Cessation; Mouth Diseases; Periodontal Diseases; Leukoplakia; Lichen Planus; Keratosis; Implant
Keywords: Smoking Cessation; Mouth Diseases; Periodontal Diseases; Leukoplakia; Keratosis; Implant; Lichen Planus
MeSH Terms: conditions — Smoking Cessation; Mouth Diseases; Periodontal Diseases; Leukoplakia; Lichen Planus; Keratosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tobacco cessation intervention (Experimental): Tobacco cessation intervention is implemented for 12 weeks. The nicotine dependence status is evaluated by the FTND (Fagerstrom Test for Nicotine Dependence) test. The point 3 or more is regarded as a moderate or high tobacco dependence and determining a cessation intervention. During the tobacco cessation intervention for the subjects, attending doctors implement standard treatments for their oral diseases. Even if participants fail to abstain from smoking, the oral treatment is continued. In case of the use of the NRTs (nicotine patch and/or gum), the investigators supply it for 2 weeks as a free of charge, and later the subjects themselves purchase it as over the counter (OTC) drugs at a pharmacy.
  Interventions: Other: Tobacco cessation intervention
- Non-tobacco cessation intervention (No Intervention): Those who do not intention to abstinence from smoking strongly and/or having less than 3 points in FTND test are allocated to non-tobacco cessation intervention group. The same treatment as the tobacco cessation intervention group is carried out for their oral diseases.

INTERVENTIONS:
Other: Tobacco cessation intervention — The nicotine dependence status is evaluated by the Fagerstrom Test for Nicotine Dependence test; those who 3 or more score are eligible for the intervention.
  During the study, attending doctors implement a tobacco cessation intervention with standard treatments for above oral diseases.
  Even if the subjects failed to abstain from smoking, the treatment is continued.
  In case of the use of the nicotine replacement therapy, The investigators supply NRTs (nicotine patch or gum) for 2 weeks as a free of charge, and later the subjects themselves purchase it as over the counter (OTC) drugs at a pharmacy.
  Arms: Tobacco cessation intervention

SUMMARY:
This study is to verify the efficacy of tobacco cessation in patients with oral diseases; periodontitis, dental implant and oral mucosal diseases by a multicenter prospective trial. Tobacco cessation intervention is implemented for 12 weeks. During the tobacco cessation intervention for the subjects, attending doctors implement standard treatments for their oral diseases. Improvement of each disease is evaluated between smoking cessation intervention group and non-cessation intervention group.

DETAILED DESCRIPTION:
It has been concluded that available evidence suggests that behavioral interventions for tobacco cessation conducted by oral health professionals incorporating an oral examination component in the dental office or community setting may increase tobacco abstinence rates among both cigarette smokers and smokeless tobacco users (Cochrane Database Syst Rev.6:CD005084.) However, efficacy of tobacco cessation for oral diseases by oral health professionals are not elucidated. There are few studies on tobacco cessation intervention by dentists but none in terms of reduction of oral diseases or further disease prevention. Association for the Japanese Academy of Maxillofacial Implants, Association for the Japanese Society of Oral and Maxillofacial Surgeons, Association for the Japanese Society of Oral Implantology, Japanese Society of Oral Medicine, Japanese Society of Periodontology, Japanese Academy of Clinical Periodontology, Japanese Society for Oral Health, Japanese Society of Dentistry for Medically Compromised Patient and Japanese Society of Oral Oncology conduct a study to verify the efficacy of tobacco cessation in patients with oral diseases; periodontitis, dental implant and oral mucosal diseases by a multicenter prospective trial.

ELIGIBILITY:
Criteria

Inclusion Criteria:

* Current smokers with periodontitis; 30% or more of the teeth where periodontal pocket depth (PPD) is 4mm or more and 3 or more sites in 6mm or more of the PPD
* Current smokers in patients about to receive implant placement
* Current smokers with oral mucosal diseases clinically diagnosed for nicotine stomatitis, oral leukoplakia, erythroplakia and oral lichen planus

Exclusion Criteria:

* Already having any cessation intervention
* Periodontitis with having anti-inflammatory drug or steroid use and have had periodontal treatment within 6 months
* Oral mucosal diseases having had surgical resections or other interventional treatments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pocket depth in peridontitis | Change from baseline at 12 months
  Pocket depth and attachment loss with or without surgical treatment
Per-implant marginal bone loss | Change from baseline at 12 months
  Per-implant marginal bone loss by a standardized X-ray photo
Size reduction of oral mucosal diseases | Change from baseline at 12 months
  Size reduction (major x minor axis /mm) at a predominant site for non-surgical group

SECONDARY OUTCOMES:
Tobacco abstinence rate | 3,6,12 and 24 months
  Biochemical validation tests confirming for quit smoking is applied for all subjects. Measurements of expired carbon monoxide (CO) where the test is available are analyzed at each period. Otherwise cotinine levels of the saliva samples are analyzed by a semi-quantitative analysis by NicAlert™.
HPV-DNA detection (p16 & 18) | pre- and post-treatment (12 months)
  The oral mucosa tissues are collected by buccal swab.

CONTACTS AND LOCATIONS:
Overall Officials: Jinichi Fukuda, PhD, DDS, Study Chair — Shin-Yurigaoka General Hospital
Locations (2):
- Japan (2):
  - Okazaki City Hospital, Okazaki, Aichi-ken
  - Shin Yurigaoka General Hospital, Kawasaki, Kanagawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440